CLINICAL TRIAL: NCT04468620
Title: A Peer-mediated Vocational Social Skills Program for Adolescents & Young Adults With Autism
Brief Title: A Peer-mediated Vocational Social Skills Program for Young Adults With Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida Gulf Coast University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-11
Record Dates: First submitted 2020-05-14; First posted 2020-07-13 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Autism Spectrum Disorder High-Functioning
Keywords: vocational rehabilitation; Mental health; social skills; employment
MeSH Terms: conditions — Psychological Well-Being; Social Skills

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ASSET Intervention (Experimental): 13-session group intervention
  Interventions: Behavioral: Assistive Soft Skills & Employment Training (ASSET)

INTERVENTIONS:
Behavioral: Assistive Soft Skills & Employment Training (ASSET) — The ASSET curriculum covers six key social skill areas: (a) Communication; (b) Networking; (c) Attitude & Enthusiasm; (d) Teamwork; (e) Problem Solving & Critical Thinking; and (f) Professionalism, as well as new content added based on our pilot findings (Mental Health; Stress Management and Self-Advocacy; and Awareness of Self & Others). The schedule includes two sessions for Communication and Professionalism, and a graduation session; thus, bringing the total number of sessions to 13. The structural elements of the training format include didactic lecture, experiential activities, group discussions, role-plays, performance feedback,and weekly take-home assignments. A key element is a social hour following each 90-minute session, in which participants practice learned skills while sharing a meal.

SUMMARY:
The Assistive Social Skills and Employment Training program (ASSET) is an occupationally-based, work-related social skills intervention, designed to address the pre-employment and mental health needs of young adults with high-functioning autism in school-to-work transition. Knowing that occupational therapy (OT) services designed to address the post-secondary transition needs of this population have been largely unexplored, and recognizing the need for OT students to gain practical experience facilitating psychosocial groups, this study seeks to: (1) evaluate program impacts on participants' psychosocial functioning and work readiness, and (2) pilot the use of OT students as group facilitators. The study will follow a mixed-methods, single group design, using questionnaires and interviews to assess skills, confidence, and psychological wellness before intervention, immediately after, and at follow-up. OT students will also be interviewed and complete pre- and post-intervention assessments of clinical self-efficacy and stress. This project supports the AOTF's objectives by: (1) building OT academic program capacity to partner with university services and the autism community to improve transition outcomes in an underserved group, (2) laying the groundwork for larger, more rigorous studies of ASSET's effectiveness, and (3) gathering pilot data to support future grant applications at the federal level.

DETAILED DESCRIPTION:
There are two specific aims of this study. First, researchers will test the effects of the ASSET Program on: (a) improving social function, work-related social skills, and self-efficacy (primary outcomes), and (b) psychological wellness (secondary outcome) using a quasi-experimental, single group, time series design. Secondly and concurrently, researchers will collect pilot data on the "near peer" mediation aspects of the intervention from the perspectives of OT students and ASSET group participants. Specifically, researchers will measure occupational therapy student facilitators' perceived stress, clinical self-efficacy, and educational value of the experience; and collect data on ASSET participants' ratings of the quality of the facilitation as delivered by occupational therapy graduate students.

Design: Using a quasi-experimental, repeated time series design, this convergent parallel mixed-methods pilot study will use quantitative data to measure change in primary and secondary outcomes, while qualitative data (session feedback forms, pre/post/follow-up interviews) will be collected in order to compare or relate themes to the quantitative findings. Building from the results of our earlier work using professional facilitators, the following two aims will be examined. Psychometric properties of instruments are available in the Appendices.

AIM 1: Evaluate the effects of the ASSET program on the social function, work-related social skills knowledge, confidence (primary outcomes) and psychological wellness (secondary outcomes) of a group of college students with HFASD immediately after the 13-week intervention delivered by graduate students and at 3-month follow-up.

Research Questions and Hypotheses:

Q1: Is ASSET associated with improvements in work-related social skills knowledge, social function, and social self-efficacy when facilitated by OTS? H1: Immediately post intervention, on average, ASSET participants will show statistically significant improvements in primary outcomes (work-related social skills knowledge, social function, and social self-efficacy).

H2: At three-month follow-up, on average, ASSET participants will show declines in primary outcomes, yet scores will remain above baseline and at statistically significant levels.

H3: Immediately post intervention, on average, ASSET participants will show clinically significant improvements in secondary mental health outcomes (anxiety and depression); however, these gains may not reach the level of statistical significance.

H4: At three-month follow-up, on average, ASSET participants will show continued improvements in secondary mental health outcomes (anxiety and depression), with improvements in anxiety reaching a level of statistical significance when compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

* 18-29 years of age
* previous diagnosis of autistic disorders, Asperger's disorder, Pervasive Developmental Disorder

Exclusion Criteria:

* no current participation in other work related social skills treatment
* no history of other neurological disorders
* no history of major mental illness (e.g., schizophrenia)

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Baseline Social Functioning | immediately pre-intervention
  Social Responsiveness System-2 (Constantino & Gruber, 2012), 65-item rating scale measuring social functioning categorized into five subscales: Social Awareness, Social Cognition, Social Communication, Social Motivation and Restricted Interests, and Repetitive Behavior. Each item is scored on a 4-point Likert-type scale, ranging from 1 (not true) to 4 (almost always true). A score decrease indicates improved functioning.
Change in Social Functioning | immediately post intervention
  Social Responsiveness System-2 (Constantino & Gruber, 2012), 65-item rating scale measuring social functioning categorized into five subscales: Social Awareness, Social Cognition, Social Communication, Social Motivation and Restricted Interests, and Repetitive Behavior. Each item is scored on a 4-point Likert-type scale, ranging from 1 (not true) to 4 (almost always true). A score decrease indicates improved functioning.
Change in Social Functioning | 85-95 days post intervention
  Social Responsiveness System-2 (Constantino & Gruber, 2012), 65-item rating scale measuring social functioning categorized into five subscales: Social Awareness, Social Cognition, Social Communication, Social Motivation and Restricted Interests, and Repetitive Behavior. Each item is scored on a 4-point Likert-type scale, ranging from 1 (not true) to 4 (almost always true). A score decrease indicates improved functioning.
Baseline General Self-efficacy | immediately pre-intervention
  The General Self-Efficacy Scale (GSE; Schwarzer and Jerusalem 1995) is a ten-item, four point Likert-type scale, ranging from 1 (not true at all) to 5 (exactly true), which measures perceived ability to cope with challenges. Higher scores indicate higher functioning.
Change in General Self-efficacy | immediately post intervention
  The General Self-Efficacy Scale (GSE; Schwarzer and Jerusalem 1995) is a ten-item, four point Likert-type scale, ranging from 1 (not true at all) to 5 (exactly true), which measures perceived ability to cope with challenges. Higher scores indicate higher functioning.
Change in General Self-efficacy | 85-95 days post intervention
  The General Self-Efficacy Scale (GSE; Schwarzer and Jerusalem 1995) is a ten-item, four point Likert-type scale, ranging from 1 (not true at all) to 5 (exactly true), which measures perceived ability to cope with challenges. Higher scores indicate higher functioning.
Baseline Perceived Empathic Self-efficacy | immediately pre-intervention
  The Perceived Empathic Self-Efficacy Scale (PESE; Caprara and Steca 2005) is a six-item self-report inventory, which measures participants' perceived ability to exercise theory of mind. The PESE uses a five-point Likert-type scale, ranging from 1 (not well at all) to 5 (very well). Higher scores indicate higher functioning.
Change in Perceived Empathic Self-efficacy | immediately post intervention
  The Perceived Empathic Self-Efficacy Scale (PESE; Caprara and Steca 2005) is a six-item self-report inventory, which measures participants' perceived ability to exercise theory of mind. The PESE uses a five-point Likert-type scale, ranging from 1 (not well at all) to 5 (very well). Higher scores indicate higher functioning.
Change in Perceived Empathic Self-efficacy | 85-95 days post intervention
  The Perceived Empathic Self-Efficacy Scale (PESE; Caprara and Steca 2005) is a six-item self-report inventory, which measures participants' perceived ability to exercise theory of mind. The PESE uses a five-point Likert-type scale, ranging from 1 (not well at all) to 5 (very well). Higher scores indicate higher functioning.
Baseline Perceived Social Self-efficacy | immediately pre-intervention
  The Perceived Social Self-Efficacy Scale (PSSE; Caprara and Steca 2005) is a five-item inventory used to measure participants' self-perceived ability to express opinions, share personal experiences, work cooperatively, and manage interpersonal conflict. Respondents rate each item on a five-point scale from 1 (not well at all) to 5 (very well). Higher scores indicate higher functioning.
Change in Perceived Social Self-efficacy | immediately post intervention
  The Perceived Social Self-Efficacy Scale (PSSE; Caprara and Steca 2005) is a five-item inventory used to measure participants' self-perceived ability to express opinions, share personal experiences, work cooperatively, and manage interpersonal conflict. Respondents rate each item on a five-point scale from 1 (not well at all) to 5 (very well). Higher scores indicate higher functioning.
Change in Perceived Social Self-efficacy | 85-95 days post intervention
  The Perceived Social Self-Efficacy Scale (PSSE; Caprara and Steca 2005) is a five-item inventory used to measure participants' self-perceived ability to express opinions, share personal experiences, work cooperatively, and manage interpersonal conflict. Respondents rate each item on a five-point scale from 1 (not well at all) to 5 (very well). Higher scores indicate higher functioning.

SECONDARY OUTCOMES:
Baseline Depression | immediately pre-intervention
  The Patient Health Questionnaire-9 (PHQ-9; Spitzer et al. 2000) is a nine-item self-report inventory used to assess depressive symptoms. The PHQ-9 uses a four-point Likert-type scale, ranging from 0 (not at all) to 3 (nearly every day) with total scores ranging from 0 to 27. Sample items include: "Little interest or pleasure in doing things," and "Feeling down, depressed, or hopeless." Lower scores indicate less symptoms.
Change in Depression | immediately post-intervention
  The Patient Health Questionnaire-9 (PHQ-9; Spitzer et al. 2000) is a nine-item self-report inventory used to assess depressive symptoms. The PHQ-9 uses a four-point Likert-type scale, ranging from 0 (not at all) to 3 (nearly every day) with total scores ranging from 0 to 27. Sample items include: "Little interest or pleasure in doing things," and "Feeling down, depressed, or hopeless." Lower scores indicate less symptoms.
Change in Depression | 85-95 days post-intervention
  The Patient Health Questionnaire-9 (PHQ-9; Spitzer et al. 2000) is a nine-item self-report inventory used to assess depressive symptoms. The PHQ-9 uses a four-point Likert-type scale, ranging from 0 (not at all) to 3 (nearly every day) with total scores ranging from 0 to 27. Sample items include: "Little interest or pleasure in doing things," and "Feeling down, depressed, or hopeless." Lower scores indicate less symptoms.
Baseline Anxiety | immediately pre-intervention
  The General Anxiety Disorder Questionnaire-7 (GAD-7; Spitzer et al., 2006) is a seven-item self-report measure used to measure anxiety. The GAD-7 uses a four-point Likert-type scale to assess frequency of symptoms, ranging from 0 (not at all) to 3 (nearly every day) with total scores range from 0 to 21. Sample items include: "Feeling nervous, anxious or on edge," and "Worrying too much about different things." Lower scores indicate less symptoms.
Changes in Anxiety | immediately post-intervention
  The General Anxiety Disorder Questionnaire-7 (GAD-7; Spitzer et al., 2006) is a seven-item self-report measure used to measure anxiety. The GAD-7 uses a four-point Likert-type scale to assess frequency of symptoms, ranging from 0 (not at all) to 3 (nearly every day) with total scores range from 0 to 21. Sample items include: "Feeling nervous, anxious or on edge," and "Worrying too much about different things." Lower scores indicate less symptoms.
Changes in Anxiety | 85-95 days post-intervention
  The General Anxiety Disorder Questionnaire-7 (GAD-7; Spitzer et al., 2006) is a seven-item self-report measure used to measure anxiety. The GAD-7 uses a four-point Likert-type scale to assess frequency of symptoms, ranging from 0 (not at all) to 3 (nearly every day) with total scores range from 0 to 21. Sample items include: "Feeling nervous, anxious or on edge," and "Worrying too much about different things." Lower scores indicate less symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Annemarie Connor, PhD, Principal Investigator — Assistant Professor
Locations (1):
- Florida Gulf Coast University, Fort Myers, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Caprara GV, Steca P, Gerbino M, Pacielloi M, Vecchio GM. Looking for adolescents' well-being: self-efficacy beliefs as determinants of positive thinking and happiness. Epidemiol Psichiatr Soc. 2006 Jan-Mar;15(1):30-43. doi: 10.1017/s1121189x00002013. PMID 16584101
- [Background] Aldridge FJ, Gibbs VM, Schmidhofer K, Williams M. Investigating the clinical usefulness of the Social Responsiveness Scale (SRS) in a tertiary level, autism spectrum disorder specific assessment clinic. J Autism Dev Disord. 2012 Feb;42(2):294-300. doi: 10.1007/s10803-011-1242-9. PMID 21516433
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Result] Connor A, Sung C, Strain A, Zeng S, Fabrizi S. Building Skills, Confidence, and Wellness: Psychosocial Effects of Soft Skills Training for Young Adults with Autism. J Autism Dev Disord. 2020 Jun;50(6):2064-2076. doi: 10.1007/s10803-019-03962-w. PMID 30879257
- [Result] Sung C, Connor A, Chen J, Lin CC, Kuo HJ, Chun J. Development, feasibility, and preliminary efficacy of an employment-related social skills intervention for young adults with high-functioning autism. Autism. 2019 Aug;23(6):1542-1553. doi: 10.1177/1362361318801345. Epub 2018 Dec 22. PMID 30582341